CLINICAL TRIAL: NCT04354103
Title: A Pilot Study to Evaluate the Effects of Atomoxetine on Impulsivity in Patients With Tourette's Syndrome
Brief Title: Atomoxetine in Patients With Tourette's Syndrome
Acronym: ATO-TS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: experimental treatment (Atomoxetine) not available
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-004455-36
Record Dates: First submitted 2020-04-07; First posted 2020-04-21 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-11

CONDITIONS: Tourette Syndrome
Keywords: Impulsivity
MeSH Terms: conditions — Tourette Syndrome; Impulsive Behavior | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with Tourette's syndrome (Experimental): Atomoxetine in Patients With Tourette's Syndrome
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — Atomoxetine

SUMMARY:
The purpose of this pilot study is to evaluate the effects of Atomoxetine, a selective noradrenaline reuptake inhibitor, on impulsivity in patients with Tourette's syndrome.

DETAILED DESCRIPTION:
High impulsivity characterizes severe forms of Tourette's syndrome, in which motor and vocal tics are associated with various neuropsychiatric disorders as compulsive disorders, difficult to manage and impairing quality of life of patients and their family. Previous preclinical study and clinical studies in attention-deficit hyperactivity disorder and Parkinson's disease demonstrate that atomoxetine, a selective noradrenaline reuptake inhibitor, improves response inhibition in high impulsive individuals. However, there is no suffisant data in Tourette's syndrome. The purpose of this pilot study is to evaluate the effects of Atomoxetine on impulsivity in 10 to 35 years old patients with Tourette's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* High impulsive patients, aged 10-35 years old, diagnosed for Tourette's syndrome as defined by the DSM-IV, never treated by Atomoxetine
* The use of effective contraception or abstinence for subjects of reproductive age
* Written informed consent

Exclusion Criteria:

* Patients with mental retardation, psychotic disorders as schizophrenia, autism spectrum disorders, chronic tics which do not respond to Tourette's syndrome criteria.
* Actual severe depression
* Allergy to one of the constituents
* Severe cardiovascular or cerebrovascular diseases, Pheochromocytoma, uncontrolled hyperthyroidism, closed angle glaucoma
* IMAO treatment discontinued less than 2 months or contra-indicated associated treatment

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Impulsive state | 8 weeks
  The primary outcome is the variation of impulsive state (%) before and after chronic administration of atomoxetine, as measured with quantitative tool (CANTAB)

SECONDARY OUTCOMES:
Cognition, anxiety, depression, severity of tics and compulsive disorders Tolerance | 8 weeks
  The secondary outcomes are the effects of Atomoxetine in cognition, anxiety, depression, severity of tics and compulsive disorders, as mesured with autoquestionnaries. The investigators also evaluate the tolerance of chronic administration of atomoxetine in patients with Tourette's syndrome.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hospices civils de Lyon, Lyon
  - AP-HP La Pitié Salpêtrière, Paris
  - CHU Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ansquer S, Belin-Rauscent A, Dugast E, Duran T, Benatru I, Mar AC, Houeto JL, Belin D. Atomoxetine decreases vulnerability to develop compulsivity in high impulsive rats. Biol Psychiatry. 2014 May 15;75(10):825-32. doi: 10.1016/j.biopsych.2013.09.031. Epub 2013 Oct 11. PMID 24252357
- [Background] Chamberlain SR, Del Campo N, Dowson J, Muller U, Clark L, Robbins TW, Sahakian BJ. Atomoxetine improved response inhibition in adults with attention deficit/hyperactivity disorder. Biol Psychiatry. 2007 Nov 1;62(9):977-84. doi: 10.1016/j.biopsych.2007.03.003. Epub 2007 Jul 17. PMID 17644072
- [Background] Kehagia AA, Housden CR, Regenthal R, Barker RA, Muller U, Rowe J, Sahakian BJ, Robbins TW. Targeting impulsivity in Parkinson's disease using atomoxetine. Brain. 2014 Jul;137(Pt 7):1986-97. doi: 10.1093/brain/awu117. Epub 2014 Jun 3. PMID 24893708
- [Background] Allen AJ, Kurlan RM, Gilbert DL, Coffey BJ, Linder SL, Lewis DW, Winner PK, Dunn DW, Dure LS, Sallee FR, Milton DR, Mintz MI, Ricardi RK, Erenberg G, Layton LL, Feldman PD, Kelsey DK, Spencer TJ. Atomoxetine treatment in children and adolescents with ADHD and comorbid tic disorders. Neurology. 2005 Dec 27;65(12):1941-9. doi: 10.1212/01.wnl.0000188869.58300.a7. PMID 16380617